CLINICAL TRIAL: NCT07109180
Title: Robot-assisted Versus Open Lateral Pancreaticojejunostomy for the Treatment of Symptomatic Chronic Pancreatitis (PANACOTTA): a Multicenter Randomized Controlled Trial
Brief Title: Robot-assisted Versus Open Lateral Pancreaticojejunostomy for the Treatment of Symptomatic Chronic Pancreatitis (PANACOTTA)
Acronym: PANACOTTA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: St. Antonius Hospital (Other); Erasmus Medical Center (Other); Maastricht University Medical Center (Other); Universitätsklinikum Hamburg-Eppendorf (Other); University Medical Center Groningen (Other); Onze Lieve Vrouwe Gasthuis (Other); Catharina Ziekenhuis Eindhoven (Other); Radboud University Medical Center (Other); Medisch Spectrum Twente (Other); Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, M.G. Besselink, M.G. Besselink, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL87297.018.24
Record Dates: First submitted 2025-07-14; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pancreatitis; Surgery; Minimally Invasive Surgical Technique; Robot Surgica; Robot Surgery; Minimally Invasive Surgery; Pancreaticojunostomy
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Who Masked: Participant
Masking Description: Patient-blinded up to post-operative day 5.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot-assisted lateral pancreaticojejunostomy (Experimental)
  Interventions: Procedure: Robot-assisted lateral pancreaticojejunostomy
- Open lateral pancreaticojejunostomy (Active Comparator)
  Interventions: Procedure: Open lateral pancreaticojejunostomy

INTERVENTIONS:
Procedure: Robot-assisted lateral pancreaticojejunostomy — Robot-assisted
  Arms: Robot-assisted lateral pancreaticojejunostomy
Procedure: Open lateral pancreaticojejunostomy — Open surgery
  Arms: Open lateral pancreaticojejunostomy

SUMMARY:
PANACOTTA is a multicenter randomized controlled trial including patients with symptomatic chronic pancreatitis and a dilated main pancreatic duct to either robot-assisted or open lateral pancreaticojejunostomy. The PANACOTTA trial will assess the post-operative quality of recovery following robot-assisted versus open lateral pancreaticojejunostomy.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Indication for (extended or partial) lateral pancreaticojejunostomy as agreed during multidisciplinary team meeting based on symptomatic chronic pancreatitis (i.e. morphine dependent pain or recurrent acute flares of pancreatitis, at least 3 episodes per year) and a dilated pancreatic duct of ≥ 5 mm, with a non-enlarged pancreatic head < 40 mm
* Confirmed CP, according to the M-ANNHEIM diagnostic Criteria24
* Eligible for both an robot-assisted and open approach
* Obtained written informed consent

Exclusion Criteria:

* Suspected or confirmed current pancreatic cancer
* ASA classification ≥ 4
* Other painful conditions aside from CP, with pain difficult to discriminate from CP pain
* Prior pancreatic surgery
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery (QoR-15) | Daily assessments on Post-operative Day 1 through Day 5 and up to time of functional recovery, defined individually per patient (maximum of 90 days from surgery).
  Primary objective: To assess post-operative mean Quality of Recovery (QoR-15) on post-operative days one through five and cumulative loss of QoR-15 until time of functional recovery of robot-assisted (RA) as compared to open lateral pancreaticojejunostomy (LPJ) in patients with symptomatic chronic pancreatitis and a dilated main pancreatic duct with a normal size pancreatic head.

CONTACTS AND LOCATIONS:
Overall Officials: M.G. Besselink, Amsterdam UMC, Principal Investigator — prof. dr.
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands